CLINICAL TRIAL: NCT03616483
Title: Collection of Specimens and Clinical Data to Create A Bio-repository for the Multiple Myeloma Program: The Indiana Myeloma Registry
Brief Title: The Indiana Myeloma Registry
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Attaya Suvannasankha, Clinical Professor of Clinical Medicine, Indiana University
Other Study IDs: IUSCC-0661
Record Dates: First submitted 2018-07-22; First posted 2018-08-06 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Plasma Cell Dyscrasias
Keywords: Multiple myeloma; Monoclonal gammopathy of undetermined significance; Plasmacytoma; Smoldering multiple myeloma
MeSH Terms: conditions — Paraproteinemias; Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Plasmacytoma; Smoldering Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, blood, bone marrow aspirate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is a non-interventional trial — This is a non-interventional trial

SUMMARY:
This is a prospective, non-interventional, observational study. The purpose of this study is to collect data and bio-specimens that will support future research

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age at the time of informed consent
2. Has been diagnosed with or is suspected to have one of the following:

   1. Monoclonal Gammopathy of Undetermined Significance (MGUS)
   2. Smoldering Multiple Myeloma
   3. Multiple Myeloma
   4. Bony or Soft Tissue Plasmacytoma
   5. Primary Amyloidosis

Exclusion Criteria:

< 18 years of age

Have not been diagnosed with one of the following:

Monoclonal Gammopathy of Undetermined Significance (MGUS) b.Smoldering Multiple Myeloma c.Multiple Myeloma d.Bony or Soft Tissue Plasmacytoma e.Primary Amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients disgnosed with one of the following:
  1. Monoclonal Gammopathy of Undetermined Significance (MGUS)
  2. Smoldering Multiple Myeloma
  3. Multiple Myeloma
  4. Bony or Soft Tissue Plasmacytoma
  5. Primary Amyloidosis
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Create a repository | 5 years
  The primary objective of this study is to provide a mechanism to store comprehensive clinical, genomic, demographic, social, environmental and quality of life data from subjects with plasma cell dyscrasias

SECONDARY OUTCOMES:
Data collection | 5 years
  To collect data related to clonal evolution, tumor microenvironment, clinical outcomes, adverse events, environmental factors and quality of life that will provide the foundation to create hypotheses for future confirmatory studies.

CONTACTS AND LOCATIONS:
Overall Officials: Attaya Suvannasankha, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No